CLINICAL TRIAL: NCT03513354
Title: Impact of a Kinesiotherapy Program on Soil and Aquatic Environment on Motor Fitness and Quality of Life of Elders. A Randomized Controlled Trial.
Brief Title: Impact of a Kinesiotherapy Program on Soil and Aquatic Environment on Motor Fitness and Quality of Life of Elders.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Federal do Rio Grande do Norte (Other)
Responsible Party: Principal Investigator, Marcelo Cardoso de Souza, Professor, PT, PhD, Universidade Federal do Rio Grande do Norte
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UFRNelders
Record Dates: First submitted 2018-04-19; First posted 2018-05-01 (Actual); Last update posted 2019-04-09 (Actual); Status verified 2019-04

CONDITIONS: Elderly
Keywords: Aging; Physical activity; Motor activity
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Intervention Model Description: 3 groups (swimming pool, soil, control group)
Who Masked: Investigator
Masking Description: blinded assessment
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control group (No Intervention): The control group did not perform any of the interventions.
- Soil group (Experimental): (2) Stretching from the lateral flexors of the cervical spine, elbow flexors and extensors, trunk lateral flexors, flexors and extensors of hip with support of 30 seconds (1x30), (3) aerobic workout through front and lateral gait walking for 20 minutes, (4) resisted exercise for upper limbs (anterior, middle and posterior deltoid, biceps, triceps) and to the lower limbs (abductors, flexors and extensors of hip and flexors and extensors knee, calf), using dumbbells and shin guards for the resistance (20 minutes), (5) balance and proprioception training through front and backward walking on mattresses, march in a straight line with one foot in front of the other, one-feet support orthostatism, touching some points marked on the ground with the toe (15 minutes)
  Interventions: Other: Soil group; Other: Pool group
- Pool group (Experimental): (2) Stretching from the lateral flexors of the cervical spine, elbow flexors and extensors, trunk lateral flexors, flexors and extensors of hip with support of 30 seconds (1x30), (3) aerobic workout through front and lateral gait walking for 20 minutes, (4) resisted exercise for upper limbs (anterior, middle and posterior deltoid, biceps, triceps) and to the lower limbs (abductors, flexors and extensors of hip and flexors and extensors knee, calf), using dumbbells and shin guards for the resistance (20 minutes), (5) balance and proprioception training through front and backward walking on mattresses, march in a straight line with one foot in front of the other, one-feet support orthostatism, touching some points marked on the ground with the toe (15 minutes)
  Interventions: Other: Soil group; Other: Pool group

INTERVENTIONS:
Other: Soil group — Exercises in soil.
  Arms: Pool group; Soil group
Other: Pool group — Exercises in pool.
  Arms: Pool group; Soil group

SUMMARY:
Introduction: Neuromotor losses are those that most affect the functionality of the elderly person. One of the preventive measures is the habit of practicing exercises regularly. Objective: To evaluate the motor fitness and the quality of life of elders before and after intervention, performed on soil and aquatic environment. Methodology: This was a randomized controlled trial, with blind evaluator and total sample of 38 elders, divided into three groups: control (n=15), soil (n=15), swimming pool (n=8). The following research instruments were used: socio-demographic data and health conditions, International Physical Activity Questionnaire (IPAQ), Mini-Mental State Examination (MMSE), Motor Scale for the Elders (MSE) and Quality of Life Questionnaire Short Form-36 (SF-36). The elders were submitted to a physiotherapeutic program during six months. Data were analyzed by statistical software Statistical Package for Social Science (SPSS 20.0). Results: When comparing motor fitness averages after intervention by study group, the soil group had higher mean values for the fine motor (p=0.021), body scheme (p=0.006), space organization (p=0.011) and general motor fitness (p=0.004) than the control group. In the quality of life, when comparing intra-group means, both intervention groups had higher averages in the general health aspect domain (p=0.001 and p=0.005 for the soil and swimming pool groups, respectively). Conclusion: This study showed that the soil group presented significantly higher means than the control group after the intervention, and the intra-group quality of life improved in both the soil as the swimming pool.

DETAILED DESCRIPTION:
The recruitment occurred in the period from October to November 2015 and the intervention was carried out from January to July 2016.

Trained evaluators applied the research instruments, the data were collected in the Faculty of Health Sciences of Trairi (FACISA). Other volunteers were responsible for conducting the intervention, other than those that evaluated.

A physiotherapeutic exercise program was applied during a period of six months, twice a week, with duration of 1 hour each session, assessing the elders before and after six months of intervention.

The same exercise program was performed, both on soil as in the swimming pool, following these steps: (1) measurement of vital signs at the beginning and at the end of the intervention: Systemic Arterial Pressure (SAP), Heart Rate (HR), Oxygen Saturation (Sp02), (2) Stretching from the lateral flexors of the cervical spine, elbow flexors and extensors, trunk lateral flexors, flexors and extensors of hip with support of 30 seconds (1x30), (3) aerobic workout through front and lateral gait walking for 20 minutes, (4) resisted exercise for upper limbs (anterior, middle and posterior deltoid, biceps, triceps) and to the lower limbs (abductors, flexors and extensors of hip and flexors and extensors knee, calf), using dumbbells and shin guards for the resistance (20 minutes), (5) balance and proprioception training through front and backward walking on mattresses, march in a straight line with one foot in front of the other, one-feet support orthostatism, touching some points marked on the ground with the toe (15 minutes).

The resisted exercise was conducted based on one maximum repetition (1MR), being used a 60% load, increasing the number of repetitions (2 repetitions) every month, starting with 2 sets of 8 repetitions in the first month, 2x10, 2x12, 2x14, 2x16 in the second, third, fourth and fifth month, respectively, ending with 2 x 18 with 60% of 1MR load and rest time of one minute between each series using dumbbells and shin guards for the resistance. In the pool, 2kg of water was used, maintaining the same series and repetitions in soil. The control group did not perform any of the interventions.

ELIGIBILITY:
Inclusion Criteria:

* (1) minimum age of 60 years, (2) presenting cognitive conditions for replying to instruments, (3) accepting and signing the ICF.

Exclusion Criteria:

* (1) presenting cognitive state suggestive of deficit according to the Mini-Mental State Examination (MMSE), (2) presenting skin infections, urinary or fecal incontinence that contraindicates the entry in the swimming pool, (3) sensory, mental and neurological changes that prevent the understanding and realization of motor testing, (4) functional limitations and/or presence of important sequels (physical disability, amputation of a member), (5) those who presented some pathology during intervention which prevented continuing the exercises.

Ages: 60 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2015-10-05 (Actual); Primary Completion 2016-05-05 (Actual); Study Completion 2016-07-05 (Actual)

PRIMARY OUTCOMES:
Mini-Mental State Examination | T0 -baseline, T6- six months (twice a week, with duration of 1 hour each session)
  Mini-Mental State Examination - with scores ranging from zero to 30 [15]. The classification of cognitive function from the MMSE score occurred as follows: 30 to 26 points - preserved cognitive functions; 26 the 24 points - change is not suggestive of deficit and 23 points or less - suggestive of cognitive deficit. The cutoff points for educational levels were the following: 18 - illiterate, 21 - elementary education and 24 - high school or higher education

SECONDARY OUTCOMES:
Motor Scale for the Elders | T0 -baseline, T6- six months (twice a week, with duration of 1 hour each session)
  Motor Scale for the Elders - validated for the Brazilian elderly population, which allows evaluating specific areas of human kinetics: fine kinetics, global kinetics, balance, body scheme, space organization and time organization [17]. Each test presents different difficulty degrees, which increases insofar as the levels advance. The results of the scores are classified into levels, as follows: far superior (130 or more), superior (120-129), high normal (110-119), average normal (90-109), low normal (80-89), low (70-79), and far low (<70)
questionnaire-Short Form 36 (SF-36) | T0 -baseline, T6- six months (twice a week, with duration of 1 hour each session)
  questionnaire-Short Form 36 (SF-36) -questionnaire with 36 items, divided into eight areas: functional capacity, physical aspects, pain, health general state, vitality, social aspects, emotional aspects, mental health and one question of comparative evaluation between current health conditions and the health conditions from the previous year [18]. Each question had a score, which were later transformed into a 0 to 100 scale, where zero corresponds to the "the worst health state" and 100, to "the best health state"

CONTACTS AND LOCATIONS:
Overall Officials: Marcelo Cardoso de Souza, PT,PhD, Principal Investigator — Adjunct Professor

IPD SHARING:
Plan to Share IPD: No
there isn't a plan to make individual participant data (IPD) available to other researchers.